CLINICAL TRIAL: NCT01577563
Title: Prevalence Study of Gastrointestinal Risk Factors in Patients With Osteoarthritis, Rheumatoid Arthritis and Ankylosing Spondylitis Receiving Treatment With Non- Steroidal Anti- Inflammatory Drugs.
Brief Title: Prevalence Study of Gastrointestinal Risk Factors in Patients With Osteoarthritis (OA), Rheumatoid Arthritis (RA) and Ankylosing Spondylitis (AS).
Acronym: RATIONAL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-PLA-XXX-2011/1
Record Dates: First submitted 2012-04-02; First posted 2012-04-16 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Osteoarthritis (OA); Rheumatoid Arthritis (RA); Ankylosing Spondylitis (AS)
Keywords: osteoarthritis (OA); rheumatoid arthritis (RA); ankylosing spondylitis (AS); gastrointestinal risk factors; NSAIDs
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
RATIONAL is a multinational, multicentre, observational, cross sectional study of adult patients in treatment with NSAID therapy for OA, RA or AS during for at least 2 weeks before study visit (at least one dose).

DETAILED DESCRIPTION:
Prevalence study of gastrointestinal risk factors in patients with osteoarthritis, rheumatoid arthritis and ankylosing spondylitis receiving treatment with non- steroidal anti- inflammatory drugs.

ELIGIBILITY:
Inclusion Criteria:

* Provision of subject informed consent.
* Female and/or male, aged > 21 years.
* Patients diagnosis with RA (ACR 1987 or ACR/EULAR 2010 criteria), OA (ACR 1986, 1990 and 1991 criteria) or AS (New York 1984 criteria or ESSG 2002 criteria) (documented in the medical record).
* Patients receiving at least one dose of NSAIDs.

Exclusion Criteria:

* Participation in any interventional study involving investigational drugs.
* Patient refuses to fill in the study questionnaires.
* Pregnant or breastfeeding women.
* Patients with active neoplastic disease in the last 5 years, except basal-cell carcinoma.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients over 21 years old, diagnosed with OA, RA or AS who are receiving at least one dose of NSAIDs for at least 2 weeks (15 days) before study visit, who attend to primary care centres, specialists offices, hospitals, private centres, urban or rural.
Sampling Method: Non-Probability Sample
Enrollment: 5383 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of subject with age above 60 years. | Up to 4 weeks.
Number of patients treated concomitantly with acetylsalicylic acid, oral corticosteroids or anticoagulants or NSAIDs. | Up to 4 weeks.
Number of patients with previous ulcer history. | Up to 4 weeks.
Number of patients with previous ulcer bleeding history. | Up to 4 weeks.
Number of patients with history of dyspepsia. | Up to 4 weeks.

SECONDARY OUTCOMES:
Descriptive profile of patients demographics: gender, ethnicity, age, educational level, professional status. | Up to 4 weeks.
Descriptive profile of medical history: nicotine use, relevant medical conditions, history peptic ulcer, chronic drug therapy related to relevant medical conditions. | Up to 4 weeks.
Descriptive profile of medical treatment with NSAIDs, ASA, PPI, DMARDs, SSRI. | Up to 4 weeks.
Descriptive profile of disease: type of rheumatic disorder: OA, RA or AS and date of first diagnosis. | Up to 4 weeks.
Descriptive profile of Health Care Resources consumption: number of hospitalizations due to the rheumatic disorder and/or GI complications. | Up to 4 weeks.
Gastrointestinal Symptoms Rating Scale (GSRS). | Up to 4 weeks.
  Rating scale for gastrointestinal symptoms in patients, consisting of five areas: reflux syndrome, abdominal pain, constipation syndrome, diarrhoea syndrome and indigestion syndrome.
Treatment Satisfaction for medication for OA patients (TSQM). | Up to 4 weeks.
  Assessment of patients' satisfaction with medication, providing scores on four scales: side effects, effectiveness, convenience and global satisfaction.
Treatment adherence (Morisky Medication Assessment Scale- MMAs-4). | Up to 4 weeks.
  A generic self-reported, medication-taking behaviour scale in which the specific health issue (e.g. rheumatic pain and dyspepsia) is inserted for the "health concern". The MMAS-4 consists of four items with a scoring scheme of "Yes" = 0 and "No" = 1. The items are added together to give a range of scores from low adherence to high adherence (0 to 4).
Patient Quality of Life (EQ-5D). | Up to 4 weeks.
  The questionnaire consists of 2 aspects: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems and severe problems.
Osteoarthritis Index capturing elements of pain and physical disability (WOMAC VA3.1). | Up to 4 weeks.
  Osteoarthritis Index, self-administered, to report health status which is designed to capture elements of pain, stiffness and physical disability in patients with OA of the knee and/or hip joints. The index consists of 24 questions (5 questions about pain, 2 on stiffness and 17 about physical function).
Health Assessment Questionnaire (HAQ). | Up to 4 weeks.
  Comprehensive measure of outcome in patients with a wide variety of rheumatic diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Citera, Rheumatologist, Study Chair — Universidad Nacional de Buenos Aires. Argentina
Locations (85):
- Argentina (22):
  - Research Site, Avellaneda, Argentina
  - Research Site, Bahía Blanca, Argentina
  - Research Site, Banfield, Argentina
  - Research Site, Campana, Argentina
  - Research Site, Capital Federal, Argentina
  - Research Site, Corrientes, Argentina
  - Research Site, La Plata, Argentina
  - Research Site, Luján, Argentina
  - Research Site, Mar del Plata, Argentina
  - Research Site, Mendoza, Argentina
  - Research Site, Olivos, Argentina
  - Research Site, Paraná, Argentina
  - Research Site, Rio Negro, Argentina
  - Research Site, Rosario, Argentina
  - Research Site, San Isidro, Argentina
  - Research Site, San Justo, Argentina
  - Research Site, San Luis, Argentina
  - Research Site, San Miguel de Tucumán, Argentina
  - Research Site, Santa Fe, Argentina
  - Research Site, Sarandi - Avellaneda, Argentina
  - Research Site, Venado Tuerto, Argentina
  - Research Site, Vicente López, Argentina
- Colombia (3):
  - Research Site, Bogotá, Colombia
  - Research Site, Bucaramanga, Colombia
  - Research Site, Cali, Colombia
- Malaysia (2):
  - Research Site, Kuala Selangor
  - Research Site, Putrajaya
- Mexico (13):
  - Research Site, Mexico City, Mexico City
  - Research Site, Aguascalientes, Mexico
  - Research Site, Boca El Rio, Mexico
  - Research Site, Cuernavaca, Mexico
  - Research Site, Durango, Mexico
  - Research Site, Guadalajara, Mexico
  - Research Site, Monterrey, Mexico
  - Research Site, Saltillo, Mexico
  - Research Site, San Luis Potosi, Mexico
  - Research Site, Tuxtla Gutierrez, Mexico
  - Research Site, Zapopan, Mexico
  - Research Site, Naucalpan, State of Mexico
  - Research Site, Toluca, State of Mexico
- Philippines (2):
  - Research Site, Davao City, Philippines
  - Research Site, Manila, Philippines
- Russia (19):
  - Research Site, Barnaul, Russia
  - Research Site, Chelyabinsk, Russia
  - Research Site, Electrostal, Russia
  - Research Site, Irkutsk, Russia
  - Research Site, Kazan', Russia
  - Research Site, Kemerovo, Russia
  - Research Site, Krasnodar, Russia
  - Research Site, Krasnoyarsk, Russia
  - Research Site, Moscow, Russia
  - Research Site, Nizhny Novgorod, Russia
  - Research Site, Novosibirsk, Russia
  - Research Site, Perm, Russia
  - Research Site, Saint Petersburg, Russia
  - Research Site, Samara, Russia
  - Research Site, Tyumen, Russia
  - Research Site, Ufa, Russia
  - Research Site, Volgograd, Russia
  - Research Site, Yaroslavl, Russia
  - Research Site, Yekaterinburg, Russia
- South Korea (11):
  - Research Site, Bucheon-si, Republic of Korea
  - Research Site, Busan, Republic of Korea
  - Research Site, Cheongju-si, Republic of Korea
  - Research Site, Daegu, Republic of Korea
  - Research Site, Hwasun-gun, Republic of Korea
  - Research Site, Incheon, Republic of Korea
  - Research Site, Jeonju, Republic of Korea
  - Research Site, Seoul, Republic of Korea
  - Research Site, Suwon, Republic of Korea
  - Research Site, Ulsan, Republic of Korea
  - Research Site, Wŏnju, Republic of Korea
- Thailand (4):
  - Research Site, Hat Yai, Thailand
  - Research Site, Klongluang, Thailand
  - Research Site, Muang, Thailand
  - Research Site, Prannok, Thailand
- Venezuela (7):
  - Research Site, Barquisimeto, Venezuela
  - Research Site, Caracas, Venezuela
  - Research Site, Maracaibo, Venezuela
  - Research Site, Maturín, Venezuela
  - Research Site, Mérida, Venezuela
  - Research Site, Porlamar, Venezuela
  - Research Site, Punto Fijo, Venezuela
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City